CLINICAL TRIAL: NCT04054427
Title: Clinical Study to Investigate Visual Performance and Patient Satisfaction After Implantation of a Trifocal Hydrophobic IOL in Patients That Underwent Refractive Surgery
Brief Title: Implantation of a Trifocal Hydrophobic IOL in Patients That Underwent Refractive Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not start study due to EC board rejection
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY1902
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular Lens; Trifocal; hydrophobic; Post refractive surgery
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOL implantation experimental (Experimental): hydrophobic, trifocal intraocular lens POD L GF
  Interventions: Device: IOL implantation experimental

INTERVENTIONS:
Device: IOL implantation experimental — Implantation of trifocal IOL POD L GF consisting of hydrophobic material

SUMMARY:
Controlled, open label, prospective Post Market Clinical Follow-Up, single-center clinical study to investigate visual performance after implantation of a trifocal IOL (PhysIOL Pod L GF) in patients that underwent refractive surgery.

DETAILED DESCRIPTION:
This clinical investigation is a controlled, open label, prospective Post Market Clinical Follow-Up, single-center clinical study whereby patients undergoing routine cataract surgery that previously underwent refractive surgery prior to being screened will have bilateral implantation of trifocal intraocular lens FineVision POD L GF (PhysIOL, Liège, Belgium).

The study purpose is to collect clinical data on visual acuity, contrast sensitivity and patient reported outcomes obtained on patients with cataracts and/or suffering from presbyopia that underwent refractive surgery prior to the IOL implantation.

The device under investigation (FineVision POD L GF) is a trifocal glistening-free hydrophobic acrylic intraocular lens (IOL) manufactured by the sponsor of this study PhysIOL sa/nv. The IOL will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

In total 28 patients will be recruited for this clinical study and receive a bilateral implantation of FineVision POD L GF intraocular lens.

Subjects participating in the trial will attend a total of 9 study visits (1 preoperative, 2 operative and 6 postoperative) over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Cataracteous eyes with no comorbidity;
* Post LASIK, post PRK/surface ablation or post RK (radial keratotomy) patients with day of refractive surgery minimum 24 months before IOL implantation;
* Calculated IOL power is within the range of the study IOLs;
* Fulfill CHRU (Centre Hospitalier Regional Universitaire) internal criteria for multifocal lenses implantation on post-refractive surgery patients.
* Male or female adults ages 45 years or older on the day of screening who have cataract(s) in one or both eyes or suffer from presbyopia;
* Clear intraocular media other than cataract;
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures;
* Signed informed consent

Exclusion Criteria:

* Age of patient < 45 years;
* Irregular topographic examination where limitation in clinical outcomes are expected.
* Patients that underwent presbyopia correcting refractive surgery (e.g. PresbyLASIK, SUPRACOR, INTRACOR)
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse;
* Subjects with AMD suspicious eyes as determined by OCT examination;
* Subjects who may be expected to require retinal laser treatment during the course of the study or at a greater risk of developing cystoid macular edema;
* Traumatic cataract;
* History or presence of macular edema;
* Concurrent or previous (within 30 days) participation in another drug or device investigation;
* Instability of keratometry or biometry measurements;
* Ocular hypertension or glaucoma;
* Significant dry eye;
* Unsuitable for study participation for any other reason, as determined by Investigator's clinical judgement (reason to be documented on the CRF).

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Monocular Best Corrected Distance Visual Acuity (CDVA) | 6 months (120-180 days) postoperative
  Statistically significant non-inferiority with POD L GF on monocular CDVA in comparison to literature data. A significance level of 0.05 will be considered statistically significant.

SECONDARY OUTCOMES:
Manifest refraction (sphere and cylinder) | Pre-OP, 1-2 days post operative, 30-60 days postoperative, 120-180 days postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2014
Pupil Size Photopic | 120-180 days postoperative
  Photopic pupil diameters are measured with a precision of at least +/-0.5 mm. For the photopic pupil diameters, eye illumination should be identical to that used for photopic contrast sensitivity testing. It is required that pupil measurements be made with an infrared pupillometer / CCD camera. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 10 minutes).
Pupil Size Mesopic | 120-180 days postoperative
  Mesopic pupil diameters are measured with a precision of at least +/-0.5 mm. For the mesopic pupil diameters, eye illumination should be identical to that used for mesopic contrast sensitivity testing. It is required that pupil measurements be made with an infrared pupillometer / CCD camera. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 10 minutes).
Uncorrected Distance Visual Acuity (UDVA) - monocular | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions
Uncorrected Distance Visual Acuity (UDVA) - binocular | 120-180 days postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Corrected Distance Visual Acuity (CDVA) - monocular | Pre-OP, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Corrected Distance Visual Acuity (CDVA) - binocular | 120-180 days postoperative
  Monocular and Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) under photopic and mesopic light conditions at 80cm distance
Uncorrected Intermediate Visual Acuity at 80cm (UIVA) - monocular | 7-14 days post operative, 30-60 days postoperative, 120-180 days postoperative
  UIVA is measured with ETDRS charts placed in 80cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Uncorrected Intermediate Visual Acuity at 80cm (UIVA) - binocular | 120-180 days postoperative
  UIVA is measured with ETDRS charts placed in 80cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 80cm (DCIVA) - monocular | 7-14 days post operative, 30-60 days postoperative, 120-180 days postoperative
  DCIVA is measured with ETDRS charts placed in 80cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 80cm (DCIVA) - binocular | 120-180 days postoperative
  DCIVA is measured with ETDRS charts placed in 80cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 80cm (DCIVA) - monocular mesopic | 120-180 days postoperative
  DCIVA is measured with ETDRS charts placed in 80cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic conditions
Uncorrected Intermediate Visual Acuity at 66cm (UIVA) - monocular | 7-14 days post operative, 30-60 days postoperative, 120-180 days postoperative
  UIVA is measured with ETDRS charts placed in 66cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Uncorrected Intermediate Visual Acuity at 66cm (UIVA) - binocular | 120-180 days postoperative
  UIVA is measured with ETDRS charts placed in 66cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 66cm (DCIVA) - monocular | 7-14 days post operative, 30-60 days postoperative, 120-180 days postoperative
  DCIVA is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 66cm (DCIVA) - binocular | 120-180 days postoperative
  DCIVA is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Distance Corrected Intermediate Visual Acuity at 66cm (DCIVA) - monocular mesopic. | 120-180 days postoperative
  DCIVA is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic conditions
Uncorrected Near Visual Acuity at 40cm (UNVA) - monocular | 7-14 days post operative, 30-60 days postoperative, 120-180 days postoperative
  UNVA is measured with ETDRS charts placed in 40cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions
Uncorrected Near Visual Acuity at 40cm (UNVA) - binocular | 120-180 days postoperative
  UNVA is measured with ETDRS charts placed in 40cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions
Distance Corrected Near Visual Acuity at 40cm (DCNVA) - monocular | 7-14 days post operative, 30-60 days postoperative, 120-180 days postoperative
  DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions
Distance Corrected Near Visual Acuity at 40cm (DCNVA) - binocular | 120-180 days postoperative
  DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions
Distance Corrected Near Visual Acuity at 40cm (DCNVA) - monocular mesopic | 120-180 days postoperative
  DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic conditions
Defocus Curve | 120-180 days postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -4.0 D to +2.0 D. This examination is performed binocularly
Binocular Contrast Sensitivity under photopic light conditions | 120-180 days postoperative
  Contrast Sensitivity under photopic light conditions using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions | 120-180 days postoperative
  Contrast Sensitivity under mesopic light conditions using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions and using a glare source | 120-180 days postoperative
  Contrast Sensitivity under mesopic light conditions with a glare source using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Patient reported outcomes: Quality of Vision Questionnaire (QoV) quality of vision | 120-180 days postoperative
  Quality of vision based on response to each question in the Quality of Vision (QoV) questionnaire. Answer is a choice of 4 options, the first being the least and the fourth being the most based on question type, i.e. "never" to "very often" or "not at all" to "severe".
Patient reported outcomes: Near Activity Visual Questionnaire (NAVQ) quality of vision | 120-180 days postoperative
  Quality of vision based on response (choice of 0-3 with 0 meaning no difficulty and 3 meaning extreme difficulty) to each question in the Near Activity Visual Questionnaire (NAVQ)
Slit lamp examination - Corneal Status | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Fundus examination with dilated pupil | Pre Op, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slit lamp examination - Signs of inflammation | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  Signs of inflammation Anterior chamber cells, Anterior chamber flare, Cystoid macular oedema, Hypopyon, and Endophthalmitis
Slit lamp examination - Pupillary block | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Pupillary block
Slit lamp examination - Retinal detachment | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Retinal detachment
Slit lamp examination - Status of anterior and posterior capsule | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Status of anterior and posterior capsule
Slit lamp examination - IOL decentration | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL decentration
Slit lamp examination - IOL tilt | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL tilt
Slit lamp examination - IOL discoloration | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL discoloration
Slit lamp examination - IOL opacity | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL opacity

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | Pre-OP, 1-2 days post operative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations. The examination is performed and documented according to the guidelines in ISO 11979-7:2018
Keratometry | Pre-OP
  Keratometric measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Biometry | Pre-OP
  Biometry measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
IOL power and target refraction | Operative (day of Surgery)
  The parameter of the implanted IOL must be recorded as well as the target refraction given by the IOL calculator. This parameter is needed to calculate the accuracy of achieving the target refraction. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus OCT | Pre-OP
  An OCT (optical coherence tomography) image will be taken at the preoperative visit to identify AMD suspicious eyes that need to be excluded from this study. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Cochener, Prof, Principal Investigator — Département d'ophtalmologie - CHU Morvan Bâtiment 4 bis

IPD SHARING:
Plan to Share IPD: No